CLINICAL TRIAL: NCT06854003
Title: A Randomized Phase 2 Study of Bendamustine, Rituximab, Cytarabine (AraC) Induction With Zanubrutinib (BRAZAN) Followed by Zanubrutinib/Rituximab +/- Sonrotoclax Maintenance in Treatment-Naïve Mantle Cell Lymphoma
Brief Title: BRAZAN: A Randomized Phase 2 Study of Bendamustine, Rituximab, Cytarabine (AraC) Induction With Zanubrutinib (BRAZAN) Followed by Zanubrutinib/Rituximab +/- Sonrotoclax Maintenance in Treatment-Naïve Mantle Cell Lymphoma
Acronym: BRAZAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christine Ryan (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor-Investigator, Christine Ryan, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-654
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Mantle Cell Lymphoma; Lymphoma
Keywords: Mantle Cell Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma | interventions — Bendamustine Hydrochloride; Rituximab; Cytarabine; zanubrutinib

STUDY DESIGN:
Intervention Model Description: Induction therapy phase followed by randomized, maintenance therapy phase. Participants will be randomized to Arms A or B, but Arm B participants requiring ramp up for Sonrotoclax, will be placed in Arm B Ramp Up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Induction Therapy (All Patients) (Experimental): Enrolled participants will complete:
  * Baseline visit with PET/CT, lymph node biopsy, and bone marrow biopsy
  * Cycles 1 through 3 (28-day cycles):
    * Days 1 - 28: Predetermined dose of Zanubrutinib 2x daily
    * Days 1 and 2: Predetermined dose of Bendamustine 1x daily
    * Day 1: Predetermined dose of Rituximab 1x daily
  * PET/CT scan
  * Cycles 4 through 6 (21-day cycles):
    * Day 1: Predetermined dose of Rituximab 1x daily
    * Days 1 and 2: Predetermined dose of Cytarabine 2x daily
  * PET/CT scan
  Participants without disease progression will proceed to randomization to either Arm A or Arm B for maintenance therapy.
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Cytarabine; Drug: Zanubrutinib
- Maintenance Arm A: Zanubrutinib + Rituximab (Experimental): Following randomization participants with a complete response to induction therapy will complete:
  * Cycles 1 - 24 (28-day cycles):
    * Days 1 through 28: Predetermined dose of Zanubrutinib 2x daily
    * Day 1 every other cycle: Predetermined dose of Rituximab 1x daily
  * PET/CT on Cycles 7, 12, 19, and at end of treatment
  * Post-treatment follow up: every 6 months. PET/CT every 12 months
  Interventions: Drug: Rituximab; Drug: Zanubrutinib
- Maintenance Arm B: Zanubrutinib + Rituximab + Sonrotoclax (Experimental): Following randomization participants with a complete response to induction therapy will complete:
  * Cycles 1 - 24 (28-day cycles):
    * Days 1 through 28: Predetermined dose of Zanubrutinib 2x daily
    * Days 1 through 28: Predetermined dose of Sonrotoclax 1x daily
    * Day 1 every other cycle: Predetermined dose of Rituximab 1x daily
  * PET/CT on Cycles 7, 12, 19, and at end of treatment
  * Post-treatment follow up: every 6 months. PET/CT every 12 months
  Interventions: Drug: Rituximab; Drug: Zanubrutinib; Drug: Sonrotoclax
- Maintenance Arm B with Sonrotoclax Ramp-Up: Zanubrutinib + Rituximab + Sonrotoclax (Experimental): Following randomization participants with an incomplete response to induction therapy will require a ramp-up initiation of sonrotoclax and will complete:
  * Cycles 1 - 24 (28-day cycles):
    * Days 1 through 28: Predetermined dose of Zanubrutinib 2x daily
    * Days 1 through 28: Predetermined dose of Sonrotoclax 1x daily
      **Cycles 1 and 2: Predetermined dose of Sonrotoclax 1x daily will be increased weekly.
    * Day 1 every other cycle: Predetermined dose of Rituximab 1x daily
  * PET/CT on Cycles 7, 12, 19, and at end of treatment
  * Post-treatment follow up: every 6 months. PET/CT every 12 months
  Interventions: Drug: Rituximab; Drug: Zanubrutinib; Drug: Sonrotoclax

INTERVENTIONS:
Drug: Bendamustine — An Alkylating agent, multi-dose vial, via intravenous (into the vein) infusion per institutional standard of care.
  Other Names: Bendamustine hydrochloride; C16H21Cl2N3O2 · HCl; Bendeka
  Arms: Induction Therapy (All Patients)
Drug: Rituximab — An Anti-CD20 antibody, single-use vials, via intravenous infusion per institutional standard of care.
  Other Names: Riabni; Rituxan; Ruxience; Truxima; ABP 798; IDEC-C2B8; PF-05280586; MabThera
Drug: Cytarabine — An Antineoplastic, single dose vial via intravenous infusion per institutional standard of care.
  Other Names: AraC
  Arms: Induction Therapy (All Patients)
Drug: Zanubrutinib — A BTK inhibitor, capsule taken orally per protocol.
  Other Names: Brukinsa; BGB-3111; C27H29N5O3
Drug: Sonrotoclax — A BCL 2 Protein Inhibitor, immediate release tablet, taken orally per protocol.
  Other Names: BGB-11417
  Arms: Maintenance Arm B with Sonrotoclax Ramp-Up: Zanubrutinib + Rituximab + Sonrotoclax; Maintenance Arm B: Zanubrutinib + Rituximab + Sonrotoclax

SUMMARY:
This study aims to evaluate the efficacy and safety of an induction regimen combining Bendamustine, Rituximab, Cytarabine (AraC), and Zanubrutinib (BRAZAN), followed by maintenance therapy with Zanubrutinib and Rituximab with or without Sonrotoclax in participants with Mantle Cell Lymphoma (MCL).

The names of the study drugs involved in this study are:

* bendamustine (a type of alkylating agent)
* rituximab (a type of monoclonal antibody)
* cytarabine (a type of antineoplastic)
* zanubrutinib (a type of kinase inhibitor)
* sonrotoclax (a type of BCL2 inhibitor)

DETAILED DESCRIPTION:
This Phase 2, multi-center, randomized study is to evaluate the efficacy and safety of an induction regimen combining Bendamustine, Rituximab, Cytarabine (AraC), and Zanubrutinib (BRAZAN), followed by maintenance therapy with Zanubrutinib and Rituximab with or without Sonrotoclax in participants with MCL. These specific maintenance therapy combinations are investigational and are being evaluated to see if the therapies may lengthen the time before MCL returns after initial therapy.

After completing induction therapy, participants will be randomized into one of two groups: Arm A: zanubrutinib + rituximab or Arm B: zanubrutinib + rituximab + sonrotoclax. Randomization means a participant is placed into a study group by chance.

The U.S. Food and Drug Administration (FDA) has approved bendamustine, cytarabine, rituximab, and zanubrutinib for the treatment of other lymphomas and/or blood cancers.

The FDA has approved rituximab as a treatment option for Mantle Cell Lymphoma (MCL).

The FDA has also approved zanubrutinib for mantle cell lymphoma, but only after trying other therapies first.

The FDA has not approved sonrotoclax as a treatment for Mantle Cell Lymphoma (MCL). However sonrotoclax works similarly to a drug called venetoclax, which is also sometimes used to treat mantle cell lymphoma. The U.S. Food and Drug Administration (FDA) has approved venetoclax for the treatment of other blood cancers.

The research study procedures include screening for eligibility, in-clinic treatment visits, electrocardiograms (ECGs), Positron Emission Tomography (PET) scans, Computerized Tomography CT) scans, blood tests, urine tests, lymph node biopsies, and bone marrow biopsies.

It is expected that about 60 people will take part in this research study.

The induction therapy will be 6 "cycles", or rounds of treatment, which will last for up to a little over 5 months. The maintenance therapy will last for up to 2 years.

* Induction phase:

  * Bendamustine/Rituximab + Zanubrutinib for 3 cycles
  * Rituximab/Cytarabine for 3 cycles
* Maintenance phase - either:

  * A) Zanubrutinib + Rituximab, or
  * B) Zanubrutinib + Sonrotoclax + Rituximab

BeiGene, Ltd., a pharmaceutical company, is also supporting this research study by providing the drugs zanubrutinib and sonrotoclax and other funding support.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of mantle cell lymphoma, with review of the diagnostic pathology specimen at one of the participating institutions. Whenever possible, the Ki67 fraction should be reported or evaluated, cytogenetics should be performed, and TP53 status should be assessed (preferably by next-generation sequencing; immunohistochemical staining would be next-preferred).
* No prior anti-lymphoma therapy, with the following exceptions:

  * Prior radiotherapy for localized disease is permitted.
  * A course of radiotherapy for urgent symptomatic disease is also permitted. Short-course systemic corticosteroids is permissible for disease control (must be < 7 days and ≤ 100mg/day of prednisone or ≤ 20mg/day of dexamethasone, or equivalent). Steroids must be discontinued prior to study treatment.
* Measurable disease, defined as ≥1 measurable nodal lesion (long axis >1.5 cm or short axis >1.0 cm) or ≥1 measurable extra-nodal lesion (long axis >1.0 cm) on PET, CT, or magnetic resonance imaging (MRI). Disease should be FDG-avid based on PET.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. (Appendix A)
* Age ≥18 years and considered a candidate for high-dose cytarabine by the treating physician.
* Adequate hematologic and organ function defined as:

  * Absolute neutrophil count ≥ 1.0 x109/L, or ≥ 0.5 x109/L if bone marrow involvement (use of growth factor support allowed).
  * Hemoglobin ≥ 8 g/dL and independent of transfusion within 7 days of screening.
  * Platelets ≥ 100 x109/L, or ≥ 50 x109/L if bone marrow involvement, and independent of transfusion within 7 days of screening.
  * Estimated CrCl ≥ 30mL/min (by Cockcroft-Gault formula or by 24-hour urine collection).
  * AST/ALT < 2.5 X institutional upper limit of normal (ULN), or < 5.0 X institutional ULN if documented liver involvement of lymphoma.
  * Total bilirubin < 2.0 X ULN (unless active hemolysis); for subjects with Gilbert's Syndrome, direct bilirubin < 1.5 X ULN.
* Patients with known infection with human immunodeficiency virus (HIV) are eligible, provided all 3 of the following are true: 1) presence of controlled disease, defined as CD4 count ≥ 200/uL and an undetectable viral load, 2) disease control has been stable on anti-retroviral therapy for at least 6 months prior to study enrollment, and 3) there are no prohibitive drug-drug interactions between study drugs and the necessary anti- retroviral therapies.
* Willingness to provide a pre-treatment tumor sample by core needle or excisional surgical biopsy. A fresh biopsy is strongly encouraged, but an archival sample is acceptable if it is collected within 90 days and without intervening treatment and the following provisions are met: 1) availability of a tumor-containing formalin-fixed, paraffin-embedded (FFPE) tissue block, 2) if the tumor containing FFPE tissue block cannot be provided in total, sections from this block should be provided that are freshly cut and mounted on positively-charged glass slides. Preferably, 25 slides should be provided; if not possible, a minimum of 15 slides is required. Exceptions to this criterion may be made with approval of the Sponsor-Investigator.
* Willingness to remain abstinent or to use two effective contraceptive methods that result in a failure rate of <1% per year from screening until at least:

  * 6 months after the last dose of bendamustine,
  * 6 months after the last dose of cytarabine,
  * 90 days after the last dose of zanubrutinib,
  * 90 days after the last dose of sonrotoclax, and/or
  * 12 months after the last dose of rituximab, whichever of the above is longest. Examples of contraceptive methods with a failure rate of <1% per year include:

    * Tubal ligation, male sterilization, hormonal implants, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
    * Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of <1% per year. Barrier methods must always be supplemented with the use of a spermicide.
    * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. In contrast, periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Known central nervous system involvement.
* Known active infection requiring systemic antimicrobial therapy at trial enrollment.
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia).
* Participants who require warfarin or other vitamin K antagonists for anticoagulation. Other anticoagulants including direct oral anticoagulants (i.e. apixaban, rivaroxaban) and low-molecular weight heparin are allowed.
* History of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusions or other medical interventions.
* History of stroke or intracranial hemorrhage within 6 months of first dose of zanubrutinib.
* History of significant or life-threatening hemorrhage within 3 months of first dose of zanubrutinib.
* History of uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia, unless these conditions are related to the underlying malignancy.
* Active hepatitis C infection. Patients with presence of HCV antibody are eligible if HCV RNA is undetectable (NOTE: the limit of detection for HCV RNA must have a sensitivity of < 15 IU/mL). Subjects who received treatment for HCV that was intended to eradicate the virus and who have an undetectable HCV RNA may participate without serial HCV RNA screening. Other patients may participate if they are willing to undergo every 3- month monitoring for HCV reactivation.
* Active hepatitis B infection. Patients with positive hepatitis B serologies with undetectable HBV DNA (NOTE: the limit of detection for HBV DNA must have a sensitivity of < 20 IU/mL) are permitted in the trial but should receive prophylactic antiviral therapy (i.e. entecavir) and undergo every 3 month HBV DNA monitoring.
* Prior history of another malignancy unless treated with curative intent and disease-free for at least 3 years at time of screening with expected low risk of recurrence during expected timeframe of study participation. Such patients should first be discussed with the Sponsor-Investigator. Additional exceptions: non-melanoma skin cancer, in situ cervical or breast cancer, or Gleason 6 prostate cancer managed with observation.
* Patients with the following cardiac conditions will be excluded:

  * New York Heart Association Class III or IV heart failure.
  * Myocardial infarction within 6 months of screening.
  * Unstable angina within 3 months prior to screening.
  * Active uncontrolled arrhythmia.
  * History of clinically significant ventricular arrhythmias within 6 months of screening (eg sustained Vtach, Vfib, torsades de pointes).
  * History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place.
  * Uncontrolled hypertension as indicated by ≥ 2 consecutive blood pressure measurements showing systolic blood pressure > 170 mm Hg and diastolic blood pressure > 105 mm Hg at screening.
* Screening 12-lead EKG showing a baseline QTcF (Fridericia's correction) > 480 msec.
* Unable to swallow capsules or disease significantly affecting gastrointestinal function, such as malabsorption syndrome.
* Participants receiving any medications or substances that are strong CYP3A inducers.

Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.

* Patients who are pregnant, breast-feeding, or intending to become pregnant during the study.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study or limit adherence to study requirements.
* Inability to comply with protocol mandated restrictions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2039-11-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) after 1-year of Maintenance Treatment | Up to 125 weeks
  CRR after maintenance treatment is defined as the proportion of participants who experienced complete response (CR) with peripheral blood (PB) MRD-negativity after 1-year of maintenance therapy.

SECONDARY OUTCOMES:
Grade 4 Treatment-Related Toxicity Rate of zanubrutinib in combination with sonrotoclax and rituximab | Up to 125 weeks
  The percentage of participants who experienced a maximum grade 4 treatment-related adverse event based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms.
Grade 4 Treatment-Related Toxicity Rate of zanubrutinib in combination with BR | Up to 125 weeks
  The percentage of participants who experienced a maximum grade 4 treatment-related adverse event based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms.
Complete Response Rate (CRR) after Maintenance Treatment in doublet arm | Up to 125 weeks
  CRR after maintenance treatment is defined as the proportion of participants who experienced complete response (CR) with PB MRD-negativity after maintenance therapy.
Complete Response Rate (CRR) after Maintenance Treatment in triplet arm | Up to 125 weeks
  CRR after maintenance treatment is defined as the proportion of participants who experienced complete response (CR) with PB MRD-negativity after maintenance therapy.
Best Overall Response (BRR) | Up to 125 weeks
  The best overall response will be the best response recorded from the start of the treatment until disease progression/recurrence.
Best Complete response (CR) rate | Up to 125 weeks
  The best CR rate will be calculated as the proportion of participants who obtained a CR at any point during study treatment.
Overall response rate (ORR) after 3 cycles of zanubrutinib + BR | Up to 125 weeks
  ORR is defined as the proportion of participants who experienced complete response (CR) or partial response (PR) after 3 cycles of zanubrutinib + BR
Complete response rate (CRR) after 3 cycles of zanubrutinib + BR | Up to 125 weeks
  CRR is defined as the proportion of participants who experienced complete response (CR) after 3 cycles of zanubrutinib + BR
Partial response rate (PRR) after 3 cycles of zanubrutinib + BR | Up to 125 weeks
  PRR is defined as the proportion of participants who experienced partial response (PR) after 3 cycles of zanubrutinib + BR
Overall response rate (ORR) after 6 cycles of BRAZAN induction | Up to 125 weeks
  ORR is defined as the proportion of participants who experienced complete response (CR) or partial response (PR) after 6 cycles of BRAZAN induction
Complete response rate (CRR) after 6 cycles of BRAZAN induction | Up to 125 weeks
  CRR is defined as the proportion of participants who experienced complete response (CR) after 6 cycles of BRAZAN induction
Partial response rate (PRR) after 6 cycles of BRAZAN induction | Up to 125 weeks
  PRR is defined as the proportion of participants who experienced partial response (PR) after 6 cycles of BRAZAN induction
Overall response rate (ORR) after the entire treatment course | Up to 125 weeks
  ORR is defined as the proportion of participants who experienced complete response (CR) or partial response (PR) after the entire treatment course
Complete response rate (CRR) after the entire treatment course | Up to 125 weeks
  CRR is defined as the proportion of participants who experienced complete response (CR) after the entire treatment course
Partial response rate (PRR) after the entire treatment course | Up to 125 weeks
  PRR is defined as the proportion of participants who experienced partial response (PR) after the entire treatment course
Overall response rate (ORR) after the entire treatment course in doublet arm | Up to 125 weeks
  ORR is defined as the proportion of participants who experienced complete response (CR) or partial response (PR) after the entire treatment course in doublet arm.
Complete response rate (CRR) after the entire treatment course in doublet arm | Up to 125 weeks
  CRR is defined as the proportion of participants who experienced complete response (CR) after the entire treatment course in doublet arm.
Partial response rate (PRR) after the entire treatment course in doublet arm | Up to 125 weeks
  PRR is defined as the proportion of participants who experienced partial response (PR) after the entire treatment course in doublet arm.
Overall response rate (ORR) after the entire treatment course in triplet arm | Up to 125 weeks
  ORR is defined as the proportion of participants who experienced complete response (CR) or partial response (PR) after the entire treatment course in triplet arm.
Complete response rate (CRR) after the entire treatment course in triplet arm | Up to 125 weeks
  CRR is defined as the proportion of participants who experienced complete response (CR) after the entire treatment course in triplet arm.
Partial response rate (PRR) after the entire treatment course in triplet arm | Up to 125 weeks
  PRR is defined as the proportion of participants who experienced partial response (PR) after the entire treatment course in triplet arm.
Duration of response (DOR) | Up to 10 years
  The duration of response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, or death due to any cause. Participants without events reported are censored at the last disease evaluation.
Duration of complete response (DOCR) | Up to 10 years
  The duration of CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented, or death due to any cause. Participants without events reported are censored at the last disease evaluation.
Duration of response (DOR) in doublet arm | Up to 10 years
  The duration of response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, or death due to any cause. Participants without events reported are censored at the last disease evaluation.
Duration of complete response (DOCR) in doublet arm | Up to 10 years
  The duration of CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented, or death due to any cause. Participants without events reported are censored at the last disease evaluation.
Duration of response (DOR) in triplet arm | Up to 10 years
  The duration of response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, or death due to any cause. Participants without events reported are censored at the last disease evaluation.
Median Duration of complete response (DOCR) in triplet arm | Up to 10 years
  The duration of CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented, or death due to any cause. Participants without events reported are censored at the last disease evaluation.
Progression free survival (PFS) | Up to 10 years
  Progression-Free Survival is defined as the time from treatment start to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Progression free survival (PFS) in doublet arm | Up to 10 years
  Progression-Free Survival is defined as the time from treatment start to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Progression free survival (PFS) in triplet arm | Up to 10 years
  Progression-Free Survival is defined as the time from treatment start to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Overall Survival (OS) | Up to 10 years
  Overall Survival is defined as the time from treatment start to death due to any cause, or censored at date last known alive.
Overall Survival (OS) in doublet arm | Up to 10 years
  Overall Survival is defined as the time from treatment start to death due to any cause, or censored at date last known alive.
Overall Survival (OS) in triplet arm | Up to 10 years
  Overall Survival is defined as the time from treatment start to death due to any cause, or censored at date last known alive.
Rate of peripheral blood (PB) MRD-negativity after 6 cycles of induction therapy | Up to 125 weeks
  Peripheral blood MRD will be measured by the clonoSEQ assay.
Rate of peripheral blood (PB) MRD-negativity after 12 cycles of maintenance treatment in doublet arm | Up to 125 weeks
  Peripheral blood MRD will be measured by the clonoSEQ assay.
Rate of peripheral blood (PB) MRD-negativity after 12 cycles of maintenance treatment in triplet arm | Up to 125 weeks
  Peripheral blood MRD will be measured by the clonoSEQ assay.
Rate of peripheral blood (PB) MRD-negativity after 24 cycles of maintenance treatment in doublet arm | Up to 125 weeks
  Peripheral blood MRD will be measured by the clonoSEQ assay.
Rate of peripheral blood (PB) MRD-negativity after 24 cycles of maintenance treatment in triplet arm | Up to 125 weeks
  Peripheral blood MRD will be measured by the clonoSEQ assay.
Best rate of peripheral blood (PB) MRD-negativity after up to 24 cycles of maintenance treatment in doublet arm | Up to 125 weeks
  Peripheral blood MRD will be measured by the clonoSEQ assay.
Best rate of peripheral blood (PB) MRD-negativity after up to 24 cycles of maintenance treatment in triplet arm | Up to 125 weeks
  Peripheral blood MRD will be measured by the clonoSEQ assay.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Ryan, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: innovation@dfci.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu